CLINICAL TRIAL: NCT06049199
Title: Assess the Effect of Speech Enhancer on Listening Effort With EEG
Brief Title: Effect of Speech Enhancer on Listening Effort With EEG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sonova AG (Industry)
Collaborators: Hoerzentrum Oldenburg (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15063
Record Dates: First submitted 2023-08-29; First posted 2023-09-22 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Listening Effort

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hearing impaired group (Experimental): The hearing impaired group will compare the reference condition (SpeechEnhancer on) with the intervention condition (SpeechEnhancer off).
  Interventions: Other: Speech Enhancer

INTERVENTIONS:
Other: Speech Enhancer — Speech Enhancer is an adaptive feature which increases the amplitude of speech signal when speech is detected. Speech Enhancer will be switched on and off for the Intervention

SUMMARY:
In previous studies, Speech Enhancer has been shown to improve Listening Effort using a subjective method. To overcome the weakness of subjective testing, this study uses an objective measurement that has shown convincing results in previous studies addressing Listening Effort.

DETAILED DESCRIPTION:
The Speech Enhancer (SE) provides better speech intelligibility for soft speech while maintaining the same sound quality for loud input level.

Better speech intelligibility may also result in less listening effort in some circumstances. So there was the hope that the SE provides better speech intelligibility and less listening effort for situation with soft speech.

The SE has already been intensely and successfully investigated in early studies.

The cognitive performance on a neurophiosiological level has already been successfully investigated in a previous studies.

ELIGIBILITY:
Inclusion Criteria:

* Experienced (minimum use duration 6 months)
* Adult (minimum age: 18 years) hearing aid users,
* Symmetrical hearing loss (difference between ears <= 10 dB for 1kHz-6kHz),
* Sensorineural hearing loss,
* Air Conduction - bone conduction gap <= 10 dB,
* Written and spoken German,
* Ability to understand instruction,
* Ability to describe listening experiences,
* Ability to attend to the appointments,
* Healthy outer ear (without previous surgical proce-dures),
* Hearing loss within the fitting ranges of the investiga-tional product,
* Informed consent as documented by signature.

Exclusion Criteria:

* Clinical contraindications deformity of the ear (closed ear canal or absence of pinna),
* Known hypersensitivity or allergy,
* Not willing to wear the hearing aid,
* Fluctuating hearing that could influence the results,
* Limited mobility and not in the position to attend all appointments,
* Inability to produce a reliable hearing test result,
* Massively limited dexterity,
* Known psychological problems,
* Known central hearing disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2023-12-22 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
EEG alpha power measured during Listening Effort Task (LET) | 10 weeks
  During the LET experiment EEG data will be recorded while participants perform the Adaptive CAtegorical Listening Effort (ACALES). Participants will be equipped with an EEG cap. A continuous EEG will be recorded while participants are performing the LET. Based on the EEG data the alpha power will be analysed offline afterwards.

SECONDARY OUTCOMES:
EEG alpha power measured during Listening Span Task (LST) | 10 weeks
  During the LST experiment EEG data will be recorded while participants perform the Working Memory Test. Participants will be equipped with an EEG cap. A continuous EEG will be recorded while participants are performing the LST. Based on the EEG data the alpha power will be analysed offline afterwards.
Listening effort (ACALES) measured during Listening Effort Task (LET) | 10 weeks
  The speech material of the ACALES is based on the German OLSA sentence matrix test. All sentences are syntactically identical and consist of five word categories (name, verb, number, adjective, and object, e.g., "Peter kauft fünf rote Blumen" [engl. "Peter buys five red flowers"]). Each trial consists of a sequence of three (different) sentences, after which participants are asked to rate their perceived listening effort on a scale via touch screen. The scale ranges from 1 (no effort) to 13 (extreme effort) based on the ACALES. These values (effort scaling units - ESCU) constitute the subjective behavioral data regarding the personal experience of listening effort.
  The ACALES is part of the LET experiment and is therefore combined with EEG recordings (see outcome 1).
Working memory measured with Listening Span Task (LST) | 10 weeks
  The material in the LST task is taken from the Basler sentence test. Half of the sentences are high predictable sentences (HP) and the other half were low predictable (LP) sentences. The participants' task is to repeat the sentence they hear and remember the last word of each sentence. After four sentences, the participants is asked to recall the final words of the last four sentences. The experimenter scores the number of correctly repeated final words after each sentence (words recognized) as well as the number of correctly recalled final words (words remembered). Based on this, a relative memory score is calculated.
  The Working Memory Test is part of the LST and is therefore combined with EEG recordings (see outcome 2).

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Vormann, Principal Investigator — Hörzentrum Oldeburg
Locations (1):
- Hörzentrum Oldenburg, Oldenburg, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wagener, K. B. (1999). Development and evaluation of a German sentence test Part II: Optimization of the Oldenburg sentence test. . Zeitschrift Fur Audiologie,, 38, 44-56.
- [Result] Krueger M, Schulte M, Brand T, Holube I. Development of an adaptive scaling method for subjective listening effort. J Acoust Soc Am. 2017 Jun;141(6):4680. doi: 10.1121/1.4986938. PMID 28679238
- [Result] Tschopp K, I. L. (1992). Die Entwicklung einer deutschen Version des SPIN-Tests (Speech Perception in Noise). In: B. Kollmeier (Hrsg): Moderne Ver-fahren der Sprachaudiometrie. . Heidelberg, Median-Verlag,, 311-329.